CLINICAL TRIAL: NCT03231501
Title: A Phase Ib, Multi-center, Open-label Study of Epitinib Succinate (HMPL-813) in Treating Patients With Glioblastoma
Brief Title: HMPL-813 in Treating Patients With Glioblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-813-00CH3
Record Dates: First submitted 2017-07-19; First posted 2017-07-27 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: This is a single arm, open label study with fixed dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): This is a single arm study. It is an open-label study. The intervention is eptinib succinate.
  Interventions: Drug: epitinib succinate

INTERVENTIONS:
Drug: epitinib succinate — This is a single-arm open label study. A subject would take 160 mg of the study medication (epitinib succinate) every day on a 28-day cycle, until he or she reaches disease progression or intolerability.

SUMMARY:
This is an open-label study, to evaluated epitinib, which is a selective epidermal growth factor receptor tyrosine kinase inhibitor (EGFR TKI), to treat glioblastoma patients with EGFR gene amplification. As epitinib could cross blood-brain barrier (BBB), inhibition of EGFR may provide a novel mechanism in treating glioblastoma.

DETAILED DESCRIPTION:
Epitinib could cross BBB and show its efficacy in brain metastasis tumors. Patients with histologically confirmed glioblastoma; standard treatment failed or no standard treatment as well as EGFR gene amplication are eligible. Patients will receive epitinib 120mg or 160mg epitinib daily. Epitinib is orally administered qd until patients reach intolerance or progression of disease. Tumor assessment takes place every 4 weeks. Simon two stage design was used, estimated making sample size of 35 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed glioblastoma
2. Standard treatment failed or no standard treatment
3. EGFR gene amplification
4. Clearly measurable lesions (according to Response Assessment in Neuro-Oncolog (RANO))
5. Age ≥ 18
6. Eastern Cooperative Oncology Group (ECOG) score ≤2

Exclusion Criteria:

1. Use of Antiepileptic drugs were used] within 2 weeks before enrollment
2. Immunotherapy, anti-angiogenesis or EGFR TKI and its downstream pathway signaling molecules and other targeted drugs within 4 weeks before enrollment; temozolomide chemotherapy, cranial radiotherapy or other systemic anti-tumor therapy within 3 weeks before enrollment
3. Previous toxic effects of anticancer therapy have not yet been recovered (defined as not restored to 0 or 1 level, except alopecia) or have not been fully recovered from previous surgery
4. Uncontrolled active infections such as acute pneumonia, Hepatitis B Virus (HBV) and so on
5. Eye disease or dry eye syndrome history
6. Positive pregnancy tested result

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 6 months
  the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period

CONTACTS AND LOCATIONS:
Overall Officials: Rongjun Liu, M.D., Study Chair — Hutchison Medipharma Ltd.
Locations (2):
- China (2):
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - The second hospital affiliated to Zhejiang University Medical School, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No